CLINICAL TRIAL: NCT06270537
Title: Multicenter Study Collecting Post-market Clinical Data on the Dominus® Stent-Graft for Treating Thoracic Aortic Diseases
Brief Title: Post-market Clinical Trial of the Dominus® Stent-Graft
Acronym: DominusPMCF
Status: Recruiting | Type: Observational
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: Dominus PMCF
Record Dates: First submitted 2024-01-09; First posted 2024-02-21 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Thoracic Aortic Dissection
Keywords: Aneurysm; Acute Aortic Syndrome; Aortic Dissection; Aortic Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aneurysm; Acute Aortic Syndrome; Aortic Dissection; Aortic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stent-Graft Dominus® Endoprosthesis — Placement of the Dominus® Stent-Graft for endovascular repair of diseases of the Thoracic Aorta

SUMMARY:
Real-world clinical trial evidence post-market, evaluating the safety and efficacy of the Dominus® StentGraft Endoprosthesis in treating thoracic aortic diseases, following the Instructions for Use

DETAILED DESCRIPTION:
The multicenter study aims to collect post-market clinical data on the Dominus® Stent-Graft in the treatment of thoracic aortic diseases. With the goal of assessing safety and efficacy, the prospective follow-up study will include 100 patients undergoing Endovascular Treatment of Thoracic Aortic Diseases, following the product's Instructions for Use

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Patients treated with the Dominus® Stent-Graft Endoprosthesis in accordance with its Instructions for Use;
3. Patient available for appropriate follow-up times for the study duration;
4. Informed patient about the nature of the study, agreeing to its provisions, and signing the informed consent.

Exclusion Criteria:

1. Patient currently participating in another clinical study of drug or medical device;
2. Life expectancy less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years and older (Adult, Older Adult )
Study Population: Patients with Thoracic Aortic Disease treated with the Dominus® Stent-Graft Endoprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Early occurrence of adverse events (Safety Outcome) | 1 month post index procedure
  Early rate Major Adverse Events (MAEs), including all-cause mortality, acute myocardial infarction (AMI), stroke, permanent paraplegia, and recent-onset renal failure (requiring dialysis).

SECONDARY OUTCOMES:
Device Success | Intraoperative
  Rate of successful introduction, navigation, and deployment of the device at the intended site
Absence of endoprosthesis fracture | 1 month and 1 year
  rate of absence of endoprosthesis fracture
Endoleak | At the end of surgery/procedure, 1 month, 6 month, 1, 2, 3, 4 and 5 years
  Rate of persistence of blood flow outside the lumen of the endoluminal graft (based on follow-up imaging). Primary endoleaks occur within 30 days post-procedure, and secondary (or late) endoleaks are detected after 30 days and subsequent to previous negative images.
Reintervention-free | At the end of surgery/procedure, 1 month, 6 month, 1, 2, 3, 4 and 5 years
  Reintervention-free rate, defined as the absence of open surgical and/or endovascular reintervention
Adverse Events | At the end of surgery/procedure, 1 month, 6 month, 1, 2, 3, 4 and 5 years
  Adverse events defined as:
  * All-cause mortality (ACM)
  * Retrograde type A dissection (RTAD)
  * Aortic rupture
  * Permanent paraplegia and paraparesis
  * Stent induced new entry tear
  * Conversation to open repair
  * Disabling stroke
  * Non-preexisting renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Edwaldo Joviliano, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo
Locations (3):
- Brazil (3):
  - Hospital Evangélico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No